CLINICAL TRIAL: NCT00948142
Title: A Phase 2, Randomized, Double-blind, Multi-center Study to Evaluate the Safety and Efficacy of CEM-102 Compared to Linezolid in the Treatment of Acute Bacterial Skin Structure Infections
Brief Title: Safety and Efficacy of CEM-102 Compared to Linezolid in Acute Bacterial Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrevus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE06-300
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Skin Diseases, Bacterial
Keywords: Acute Bacterial Skin and Skin Struction Infections; Bacterial Skin Diseases; Staphylococcal Skin Infections; MRSA
MeSH Terms: conditions — Skin Diseases, Bacterial; Staphylococcal Skin Infections | interventions — Fusidic Acid; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Linezolid (Active Comparator): 600 mg BID
  Interventions: Drug: Linezolid
- CEM-102 Regimen A (Experimental)
  Interventions: Drug: CEM-102
- CEM-102 Regimen B (Experimental)
  Interventions: Drug: CEM-102

INTERVENTIONS:
Drug: CEM-102 — 600 mg BID oral tablets for 10-14 days
  Other Names: fusidic acid
  Arms: CEM-102 Regimen A
Drug: Linezolid — 600 mg BID oral tablets
  Other Names: Zyvox
  Arms: Linezolid
Drug: CEM-102 — 1500 mg BID oral tablets on Day 1 followed by 600 mg BID oral tablets for a total of 10-14 days
  Other Names: fusidic acid
  Arms: CEM-102 Regimen B

SUMMARY:
The purpose of this study is to determine the safety and efficacy of CEM-102 compared to Linezolid in the treatment of acute bacterial skin structure infections (ABSSIs).

DETAILED DESCRIPTION:
ABSSIs are common and affect all age groups. In recent years, ABSSIs caused by multi-drug resistant pathogens, especially methicillin-resistant Staphylococcus aureus (MRSA) have become more common. There is an urgent need for additional antibacterial drugs with modes of action different from those currently available. CEM-102 is one such agent with excellent activity against S. aureus, including MRSA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute bacterial skin-structure infection (ABSSI) of no more than 7 days duration which was suspected or proven to be caused, at least in part, by a gram-positive pathogen.
* Eligible infections included cellulitis measuring at least 10 cm length and width or 100 cm squared, with or without a focal abscess, and surgical or traumatic wound infections
* Infection which in the opinion of the investigator will require 10-14 days of antibacterial therapy.
* Have at least 3 of the following local and/or systemic symptoms and/or signs of infection: purulent or seropurulent drainage/discharge, erythema, fluctuance, heat/localized warmth, pain/tenderness to palpation, swelling/induration, regional lymph node swelling or tenderness, temperature >=100.4 degree F, increased white blood cell count, or bandemia.
* Must not have received treatment with another systemic antibiotic for the current ABSSI.

Exclusion Criteria:

* Superficial skin structure infections such as folliculitis, carbuncles, furunculosis, cutaneous abscesses, and simple cellulitis.
* Infections involving burns, human or animal bites, or chronic diabetic foot ulcers.
* Suspected polymicrobial infection involving Pseudomonas aeruginosa
* Anticipated need for >14 days of antibiotic therapy.
* Infections complicated by the presence of prosthetic materials that will not be removed, such as permanent cardiac pacemaker battery packs, mesh, or joint replacement prosthesis.
* Known significant renal, hepatic, or hematologic impairment.
* Received prior potentially effective antimicrobial therapy for the acute bacterial skin and skin structure infection, unless they were failing therapy after 48 hours or had a gram-positive pathogen non-susceptible to prior therapy identified as a causative pathogen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Clinical Success at Test of Cure (TOC) for the intent-to-treat (ITT) population | 7 to 14 days after the last dose of study drug
  Meets the following definition for clinical success: continued complete resolution of the signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required
Clinical Success at Test of Cure (TOC) for the clinically evaluable (CE) population | 7 to 14 days after the last dose of study drug
  Meets the following definition for clinical success: continued complete resolution of the signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required

SECONDARY OUTCOMES:
Clinical Success at end of treatment (EOT) for the intent-to-treat (ITT) population | 10-14 days of study drug
  Meets the following definition for clinical success: Complete resolution of the signs and symptoms of the ABSSI and no further study drug therapy is required.
Clinical Success at the test of cure (TOC) in the microbiological intent-to-treat (MITT) and population | 7 to 14 days after the last dose of study drug
  Meets the following definition for clinical success: Complete resolution of the signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required.
Clinical Success at the end of treatment (EOT) for the Clinically evaluable (CE) population | 10-14 days of study drug
  Meets the following definition for clinical success: complete resolution of the signs and symptoms of the ABSSI and no further study drug therapy is required.
Clinical success at the end of treatment (EOT) for the microbiological intent-to-treat (MITT) population | 10-14 days of study drug
  Meets the following definition for clinical success at the end of treatment: complete resolutoin of the signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required
Clinical Success at end of treatment (EOT) for the microbiologically evaluable (ME) population | 10-14 days of study drug
  Meets the following definition for clinical success: complete resolution of signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required.
Clinical Success at test of cure (TOC) for the microbiologically evaluable (ME) population | 7-14 days after the last dose of study drug
  Meets the following definition of clinical success: continued complete resolution of the signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required.
Clinical success at the test of cure (TOC) by baseline pathogen for the microbiological intent-to-treat (MITT) population | 7-14 days after the last dose of study drug
  Meets the following definition for clinical success: continued complete resolution of the signs and symptoms of the ABSSI and no additonal systemic antibacterial therapy is required
Clinical success at test of cure (TOC) by baseline pathogen for the microbiologically evaluable (ME) population | 7 to 14 days after the last dose of study drug
  Meets the following definition for clinical success: continued complete resolution of the signs and symptoms of the ABSSI and no additional systemic antibacterial therapy is required
By-pathogen microbiological success at test of cure (TOC) for the microbiological intent-to-treat (MITT) population | 7-14 days after the last dose of study drug
  Successful responses included:
  eradication: the basline causative pathogen was absent from the culture(s) presumed eradication: the patient's clincial response was success, and no culture available.
By-pathogen microbiological success at test of cure (TOC) for the microbiologically evaluable (ME) population | 7-14 days after the last dose of study drug
  Successful responses included:
  eradication: the basline causative pathogen was absent from the culture(s) presumed eradication: the patient's clincial response was success, and no culture available.
By-patient microbiological success at test of cure (TOC) for the microbiological intent-to-treat (MITT) population | 7-14 days after the last dose of study drug
  Successful responses included:
  eradication: the baseline causative organisms have a response of eradication. presumed eradication: all baseline causative organism(s) have a response of presumed eradication combined eradication/presumed eradication: in cases where baseline causative organisms were from a blood and an ABSSI culture
By-patient microbiological success at test of cure (TOC) for the microbiologically evaluable (ME) population | 7-14 days after the last dose of study drug
  Successful responses included:
  eradication: the baseline causative organisms have a response of eradication. presumed eradication: all baseline causative organism(s) have a response of presumed eradication combined eradication/presumed eradication: in cases where baseline causative organisms were from a blood and an ABSSI culture

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Chula Vista, California
  - La Mesa, California
  - Los Angeles, California
  - Oceanside, California
  - Oxnard, California
  - Pasadena, California
  - Santa Ana, California
  - Torrance, California
  - Columbus, Georgia
  - Savannah, Georgia
  - Springfield, Illinois
  - Detroit, Michigan
  - Butte, Montana
  - Somers Point, New Jersey
  - Akron, Ohio

REFERENCES:
- [Derived] Craft JC, Moriarty SR, Clark K, Scott D, Degenhardt TP, Still JG, Corey GR, Das A, Fernandes P. A randomized, double-blind phase 2 study comparing the efficacy and safety of an oral fusidic acid loading-dose regimen to oral linezolid for the treatment of acute bacterial skin and skin structure infections. Clin Infect Dis. 2011 Jun;52 Suppl 7:S520-6. doi: 10.1093/cid/cir167. PMID 21546629